CLINICAL TRIAL: NCT04010565
Title: Effect of a Black Garlic Extract With Greater Concentration of Bioactive Compounds and Lower Content in Undesired Compounds on Cholesterol LDL Levels. Chronic, Randomized, Crossover, Controled and Double Blind Study
Brief Title: Effect of a Black Garlic Extract on Cholesterol LDL Levels
Acronym: ESACTIVO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technological Centre of Nutrition and Health, Spain (Other)
Collaborators: Fundació Eurecat (Other); Hospital Universitari Sant Joan de Reus (Other); University Rovira i Virgili (Other); Pharmactive Biotech Products S.L. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ESACTIVO
Record Dates: First submitted 2019-07-03; First posted 2019-07-08 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Cardiovascular Diseases
Keywords: Cholesterol LDL; Black garlic extract; S-allyl cysteine
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The consumption of SANE and placebo will be in the form of tablets with the same appearance, of 550 mg / tablet, guaranteeing that the study is blind both for the researchers of the project and for the participants (double blind).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extract of aged black garlic (Experimental): Participants will consume a tablet of 550 mg daily with 250 mg of aged black garlic extract and 300 mg of excipients (microcrystaline cellulose 90 mg; dicalcium phosphate 157 mg; crosscamellose sodium 10 mg; magnesium stearate 7 mg; sodium alignate 3.06 mg; stearic acid 0.03 mg; oleic acid 1.54 mg; medium chain triglycerides 2.80 mg; ethylcellulose 13.17 mg; hydroxypropylcellulose 4.86 mg; hydroxypropylmethylcellulose 4.86 mg; talcum 2.88 mg; titanium dioxide 1.80 mg; vanilla aroma 1.00 mg) .
  Interventions: Dietary Supplement: Aged black garlic extract
- Placebo (Placebo Comparator): Participants will consume a tablet of 550 mg daily with 550 mg of excipients (microcrystaline cellulose 342.5 mg; dicalcium phosphate 154.5 mg; crosscamellose sodium 10 mg; magnesium stearate 7 mg; sodium alignate 3.06 mg; stearic acid 0.03 mg; oleic acid 1.54 mg; medium chain triglycerides 2.80 mg; ethylcellulose 13.17 mg; hydroxypropylcellulose 4.86 mg; hydroxypropylmethylcellulose 4.86 mg; talcum 2.88 mg; titanium dioxide 1.80 mg; vanilla aroma 1.00 mg).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Aged black garlic extract — Participants will intake a tablet with 250 mg of a aged black garlic extract with higher concentration of bioactive compounds S-allyl cysteine and alliin, and minor unwanted compounds such as simple sugars and furfural derivatives.
  In addition, during the course of the study, participants will be urged to follow dietary guidelines according to a heart-healthy diet established by nutritionists and that they will adhere to European guidelines for the treatment of dyslipidemias.
  Arms: Extract of aged black garlic
Dietary Supplement: Placebo — Participants will intake a tablet with 250 mg of microcrystalline cellulose. In addition, during the course of the study, participants will be urged to follow dietary guidelines according to a heart-healthy diet established by nutritionists and that they will adhere to European guidelines for the treatment of dyslipidemias.
  Arms: Placebo

SUMMARY:
One of the most characteristic components of the Mediterranean diet is garlic (Allium sativum L.), food to which has been attributed protective properties against cardiovascular diseases (CVD). Recently, several methods of garlic processing have been developed to obtain derivatives with milder organoleptic characteristics and a longer shelf life than habitual garlic derivates. One of these strategies is the aging of the garlic by high temperatures treatment that eliminates the taste and characteristic odor of garlic and gives it a dark color, a sweet taste and a slimy texture. Because the changes in the visual and organoleptic characteristics, the garlic obtained by aging at high temperatures is named black garlic.

Interestingly, these modifications translate into an increase in their antioxidant power and their protective capacity against the development of CVDs, mainly due to the formation of melanoidins and to the content of organosulfur derivatives of cysteine compounds, such as S-allyl-cysteine (SAC) and alliin.

Hypothesis of the study: The daily administration of a new extract of aged black garlic (SANE), with a higher concentration of bioactive compounds and lower unwanted compounds will lower cholesterol levels of low density lipoproteins (LDL-c), and will produce favorable changes on other markers of cardiovascular risk in individuals with moderate hypercholesterolemia.

Each 250 mg of SANE contains 0.5% in SAC, which will mean an amount of 1.25 mg of SAC per day, about 5 times more than SAC levels present in many of the black garlic products marketed.

The main objective was to evaluate the effect of the daily intake of a SANE with a higher concentration of bioactive compounds, SAC and alliin, and minor unwanted compounds such as simple sugars and furfural derivatives, in combination with dietary recommendations, on LDL-c levels in individuals with moderate hypercholesterolemia.

DETAILED DESCRIPTION:
Chronic, randomized, crossover, placebo-controlled and double-blind nutritional intervention trial.

The 60 participants in the study will be randomly divided into two groups of 30 participants, as they begin the study taking the SANE or placebo for 6 weeks.

At the end of study week 6, when the first treatment is finished, a 3-week washout period will be carried out, and then the treatment that will take place during another 6 weeks will be exchanged. Total study duration of 15 weeks.

The dose of SANE will be 250 mg daily, presented in a tablet of 550 mg / unit. The placebo will be microcrystalline cellulose. The consumption of SANE and placebo will be in the form of tablets with the same appearance, of 550 mg / tablet, guaranteeing that the study is blind both for the researchers of the project and for the participants (double blind).

The tablets will be presented in recipients of 45 units, so that with one recipient the participants will be able to carry out the entire intervention for each of the products.

Adverse effects will be controlled: body odor, halitosis, flatulence, nausea, abdominal distension, reflux and allergic reactions.

During the study, volunteers will perform 7 visits, according to the cross-type study design.

* a pre-selection visit (to check inclusion / exclusion criteria) (V0) and, in case of meeting the inclusion criteria,
* three study visits during the consumption of SANE, which will take place in weeks 1 (start of the study), 3 and 6 (end point) (V1, V2, V3).
* three study visits during the consumption of the placebo, which will take place in weeks 1 (start of the study), 3 and 6 (end point) (V4, V5, V6).

In all the visits the participants must present themselves in fasting conditions of 8 hours to obtain blood. In addition, at each visit (except in the case of V0) a questionnaire will be conducted to determine the presence / absence of adverse effects.

Main variable: LDL-c concentrations.

Secondary variables:

* Measures of body composition (in all study visits, V0-V6):
* Body weight.
* Height.
* Body mass index (BMI) (Kg / m2).
* Waist circumference.
* Blood pressure (in all study visits, V0-V6):
* Systolic blood pressure (SBP).
* Diastolic blood pressure (DBP).
* Parameters in plasma:
* Total cholesterol, High density lipoproteins cholesterol (HDL-c) and triglycerides (TG) (in all study visits, V0-V6).
* From these values the atherogenic indices (AIs) will be calculated:
* Total cholesterol / HDL-c;
* LDL-c / HDL-c
* Plasma atherogenic index, which combines the values of triglycerides and HDL-c, calculated as the logarithm of the TG / HDL-c ratio, which is considered a good indirect indicator of the size of the LDL-c particles and of the subclinical atherosclerosis.
* Glucose (in all the visits of the study, V0-V6).
* Insulin and Non esterified free fatty acids (NEFAs) (at the beginning and end of the study period visits with each of the two products (SANE or placebo).
* From the glucose and insulin values, the Homeostatic Model Assessment for insulin resistance index (HOMA-IR) and the revised-Quantitative insulin sensitivity index (R-QUICKI) will be calculated.
* The pro-inflammatory cytokines Monocyte chemoattractant protein 1 (MCP-1), Interleukin 6 (IL-6) and (Tumor necrosis factor alpha (TNF-α) (at the beginning and end of the study period visits with each of the two products (SANE or placebo).
* Apolipoprotein (Apo) B, a protein present in the potentially atherogenic particles present in plasma and that reflects the number of particles that contain cholesterol and triglycerides (in the visits of the beginning and end of the study period with each of the two products (SANE or placebo).
* Apo A1, the major protein present in HDL-c and that initiates the reverse transport of cholesterol (in the visits of the beginning and end of the study period with each of the two products (SANE or placebo).
* Based on the ApoB and ApoA1 values, the Apo B / Apo A1 ratio will be calculated as an indicator of cardiovascular disease risk. This ratio reflects the balance between proatherogenic and CVD protective particles.
* Oxidized LDL-c (oxLDL) (at the beginning and end of the study period visits with each of the two products (SANE or placebo).
* Phospholipid transfer protein (PLTP) (at the start and end visits of the study period with each of the two products (SANE or placebo).

ELIGIBILITY:
Inclusion Criteria:

1. Men and women over 18 years of age.
2. Fasting serum LDL-c concentration ≥ 115 mg/dL.
3. Sign the informed consent.

Exclusion Criteria:

1. BMI ≥ 35 kg/m^2
2. LDL-c serum levels <115 mg/dL
3. Serum glucose levels higher than 126 mg/dL
4. Take supplements or multivitamin supplements or phytotherapeutic products that interfere with the treatment under study up to 30 days before the start of the study.
5. Be a smoker
6. Follow a hypocaloric diet and/or pharmacological treatment for weight loss.
7. Anti-hypertensive treatment.
8. Presenting anemia (hemoglobin ≤ 13 g/dL in men and ≤ 12 g/dL in women).
9. Present some chronic gastrointestinal disease.
10. Present some chronic disease in clinical manifestation.
11. Being pregnant or intending to become pregnant.
12. Be in breastfeeding period.
13. Participate in or have participated in a clinical trial or nutritional intervention study in the last 30 days prior to inclusion in the study.
14. Being unable to follow the study guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
LDL-c levels | At week 1, week 3 and week 6 for each of the two treatments (SANE and placebo).
  Serum LDL-c levels will be measured by standardized methods in Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain).

SECONDARY OUTCOMES:
Measures of body weight | At week 1, week 3 and week 6 for each of the two treatments (SANE and placebo).
  Body weight measured by TANITA SC330.
Measures of height | At week 1, week 3 and week 6 for each of the two treatments (SANE and placebo).
  Height measured by standardized methods.
Measures of BMI | At week 1 for each of the two treatments (SANE and placebo).
  Weight and height will be combined to report BMI in kg/m^2.
Measures of waist circumference | At week 1, week 3 and week 6 for each of the two treatments (SANE and placebo).
  Waist circumference using a measuring tape.
Bood pressure (measured in mmHg) | At week 1, week 3 and week 6 for each of the two treatments (SANE and placebo).
  Systolic and diastolic blood pressure will be measured twice after 2-5 minutes of patient respite, seated, with one-minute interval in between, using an automatic sphygmomanometer (OMRON HEM-907; Peroxfarma, Barcelona, Spain).
Lipid metabolism | At week 1, week 3 and week 6 for each of the two treatments (SANE and placebo).
  Total cholesterol, HDL-c, TG, NEFAs, Apo B and Apo A1 plasma levels will be measured by standardized methods in Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain). oxLDL, PLTP plasma levels will be measured by human ELISA kits.
Glucose metabolism | At week 1, week 3 and week 6 for each of the two treatments (SANE and placebo).
  Glucose and insulin plasma levels will be measured by standardized methods in Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain).
Inflammation | At week 1, week 3 and week 6 for each of the two treatments (SANE and placebo).
  IL-6 plasma levels will be measured by standardized methods in Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain). MCP-1 and TNF alpha will be measured by human ELISA kits.

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Solà, Dr, Principal Investigator — Centro Tecnológico de Nutrición y Salud (Eurecat_Reus). Reus, Tarragona, Spain.
Locations (1):
- Centro Tecnológico de Nutrición y Salud (Eurecat-Reus), Reus, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Technological Centre of Nutrition and Health. Eurecat_Reus. — http://eurecat.org